CLINICAL TRIAL: NCT00901901
Title: A Phase III Randomized, Placebo Controlled, Double Blind Trial of Sorafenib Plus Erlotinib vs. Sorafenib Plus Placebo as First Line Systemic Treatment for Hepatocellular Carcinoma (HCC)
Brief Title: Nexavar-Tarceva Combination Therapy for First Line Treatment of Patients Diagnosed With Hepatocellular Carcinoma
Acronym: SEARCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12917; 2008-006021-14 (EudraCT Number)
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Sorafenib (Nexavar); Erlotinib (Tarceva); First Line; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) (Experimental): Participants received sorafenib 400 mg twice daily (bid) and erlotinib 150 mg tablet once daily (qd)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Erlotinib (Tarceva)
- Sorafenib (Nexavar, BAY43-9006) + Placebo (Active Comparator): Participants received sorafenib 400 mg twice daily (bid) and matching erlotinib placebo 150 mg tablet once daily (qd)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 400 mg twice daily
Drug: Erlotinib (Tarceva) — Erlotinib 150 mg once daily
  Arms: Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva)
Drug: Placebo — Matching erlotinib placebo 150 mg once daily
  Arms: Sorafenib (Nexavar, BAY43-9006) + Placebo

SUMMARY:
This is a randomized trial to evaluate the clinical benefit of sorafenib 400 mg twice daily and erlotinib 150 mg once a day versus sorafenib 400 mg twice daily and placebo erlotinib once daily in subjects with unresectable advanced or metastatic Child-Pugh A HCC. Patients who are candidates for potentially curative intervention (i.e. surgical resection or local ablation) are not eligible for this study.

DETAILED DESCRIPTION:
European quality of life scale (5 dimensions) (EQ-5D)

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients who have a life expectancy of at least 12 weeks
* Patients with histological or cytologically documented HCC
* Patients must have at least one tumor lesion that meets both of the following criteria:

  * The lesion can be accurately measured in at least one dimension according to response evaluation criteria in solid tumors (RECIST)
  * The lesion has not been previously treated with local therapy
* Patients who have an ECOG PS (Eastern Cooperative Oncology Group Performance Status) of 0 or 1
* Cirrhotic status of Child-Pugh class A.
* Patients who give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time.

Exclusion Criteria:

* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) class 2; active coronary artery disease (CAD); cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin), or uncontrolled hypertension. Myocardial infarction more than 6 months prior to study entry is permitted.
* Abnormalities of the cornea based on history (e.g. dry eye syndrome, Sogren's syndrome) including congenital abnormality (e.g. Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g. fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test).
* History of interstitial lung disease (ILD).
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Previous treatment with yttrium-90 spheres
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2009-05-21 (Actual); Primary Completion 2012-04-17 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (115):
- United States (22):
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Maywood, Illinois
  - Westwood, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - New York, New York
  - Rochester, New York
  - Valhalla, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
- Australia (6):
  - Randwick, New South Wales
  - Brisbane, Queensland
  - Herston, Queensland
  - Clayton, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Vienna, Austria
- Belgium (7):
  - Bruxelles - Brussel
  - Edegem
  - Ghent
  - Kortrijk
  - La Louvière
  - Leuven
  - Liège
- Brazil (5):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
  - São Paulo
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Canada (2):
  - Edmonton, Alberta
  - Montreal, Quebec
- Santiago, Chile
- China (4):
  - Guangzhou, Guangdong
  - Nanjing, Jiangsu
  - Hangzhou, Zhejiang
  - Beijing
- Colombia (2):
  - Floridablanca
  - Medellín
- France (11):
  - Bordeaux
  - Clichy
  - Créteil
  - La Roche-sur-Yon
  - Lille
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (11):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Regensburg, Bavaria
  - Frankfurt am Main, Hesse
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Berlin
- Greece (3):
  - Athens
  - Larissa
  - Thessaloniki
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Israel (5):
  - Beersheba
  - Haifa
  - Petah Tikva
  - Rehovot
  - Zrifin
- Milan, Lombardy, Italy
- New Zealand (3):
  - Auckland
  - Christchurch
  - Wellington South
- Lima, Peru
- Poland (4):
  - Bydgoszcz
  - Gdansk
  - Gliwice
  - Warsaw
- Russia (3):
  - Barnaul
  - Moscow
  - Nizhny Novgorod
- Singapore, Singapore
- South Africa (2):
  - Johannesburg, Gauteng
  - Cape Town, Western Cape
- South Korea (2):
  - Goyang-si, Gyeonggido
  - Seoul
- Spain (6):
  - L'Hospitalet de Llobregat, Barcelona
  - Barcelona
  - Lugo
  - Madrid
  - Santander
  - Valencia
- Taiwan (3):
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (4):
  - Sheffield, South Yorkshire
  - Glasgow
  - London
  - Newcastle upon Tyne

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 128 study centers in 26 countries in North America, South America, Europe, Africa, and Asia.
Pre-assignment Details: Of the 962 screened participants, 242 were screen failures and were excluded from participated in the study. A total of 720 participants were randomized to study arms: 358 participants in the sorafenib + placebo group and 362 participants in the sorafenib + erlotinib group.
Period: Treatment Period
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY43-9006) + Placebo
Started | 362 | 358
Participants Received Treatment | 362 | 355
Completed | 193 | 181
Not Completed | 169 | 177
Not completed — Adverse Event | 120 | 128
Not completed — Withdrawal by Subject | 26 | 24
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 3 | 5
Not completed — Noncompliance with study medication | 4 | 1
Not completed — Missing | 1 | 0
Not completed — Never treated | 0 | 3
Not completed — Protocol driven decision point | 0 | 2
Not completed — Study terminated by sponsor | 2 | 0
Not completed — Protocol Violation | 5 | 9
Not completed — Switch to commercial drug | 1 | 1
Not completed — Transfer to treatment continuation study | 5 | 2
Period: Follow-up Period
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY43-9006) + Placebo
Started | 340 | 341
Completed | 0 | 0
Not Completed | 340 | 341
Not completed — Death | 181 | 208
Not completed — Protocol driven decision point | 47 | 36
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 12 | 8
Not completed — Missing | 94 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY43-9006) + Placebo | Total
Number analyzed (Participants) | 362 | 358 | 720
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (11.8) | 59.5 (13.0) | 59.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 139
  Male | 295 | 286 | 581
Smoking status [Count of Participants; unit: Participants]
  non-smoker | 112 | 107 | 219
  former smoker | 132 | 128 | 260
  current smoker | 118 | 123 | 241
ECOG stratification group [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) grade 0 = fully active; grade 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    0 | 222 | 216 | 438
    1 | 140 | 142 | 282
Macroscopic vascular invasion [Count of Participants; unit: Participants]
  Yes | 138 | 153 | 291
  No | 224 | 205 | 429
Extrahepatic spread [Count of Participants; unit: Participants]
  Yes | 205 | 219 | 424
  No | 157 | 139 | 296

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from date of randomization to death due to any cause.
Time Frame: From randomization of the first patient until 34 months or date of death of any cause whichever came first
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Days | 289 [250 to 321] | 259 [226 to 322]

2. Secondary Outcome: Time to Radiological Tumor Progression (TTP)
Description: TTP was the time from randomization to radiological tumor progression. Participants without radiological tumor progression at the time of analysis were censored at their last date of tumor evaluation. Progressive disease (PD) was defined using Response Evaluation Criteria in Solid Tumors (RECIST version 1.0), as at least a 20% increase in the sum of longest diameter (LD) of measured lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Appearance of new lesions also constituted PD.
Time Frame: From randomization of the first participant until 34 months later (cut-off date), assessed every 6 weeks
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva): Participants received sorafenib 400 mg twice daily (bid) and erlotinib 150 mg tablet once daily (qd)
- Sorafenib (Nexavar, BAY 43-9006) + Placebo: Participants received sorafenib 400 mg twice daily (bid) and matching erlotinib placebo 150 mg tablet once daily (qd)
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Days | 97 [82 to 126] | 122 [88 to 136]

3. Secondary Outcome: Disease Control
Description: Disease control was defined as the number of participants who had a best response rating of complete response (CR), partial response (PR), or stable disease (SD) according to RECIST assessed by magnetic resonance imaging (MRI) that was confirmed at least 28 days from the first demonstration of that rating. CR: disappearance of all clinical and radiological evidence of target and non-target tumors. PR: at least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD. SD: steady state of disease. Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: From randomization of the first participant until 34 months later (cut-off date), assessed every 6 weeks
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Participants | 159 | 188

4. Secondary Outcome: Health-related Quality of Life and Utility Values as Measured by EQ-5D - Index
Description: The European quality of life scale (5 dimensions) (EQ-5D) questionnaire was given to the participants at each visit. The EQ-5D questionnaire consisted of 5 ordinal categorical responses (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The scores for the EQ-5D dimensions are assigned according to the level of problems reported (1 'no problems'; 2 'some problems'; 3 'extreme problems'). The 5 health dimensions are summarized into a single score, the EQ-5D index score. The EQ-5D index score has a range of 0 and 1 with 0 representing death and 1 representing perfect health.
Time Frame: The EQ-5D was administered at the beginning of the visit prior to seeing the investigator. Questionnaires were to be completed every 6 weeks (Day 1 of each cycle) for subsequent cycles and at the end of treatment visit.
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Scores on a scale
  cycle1 | 0.777 [0.760 to 0.795] | 0.774 [0.757 to 0.790]
  cycle2 | 0.753 [0.735 to 0.771] | 0.749 [0.732 to 0.766]
  cycle3 | 0.728 [0.708 to 0.748] | 0.724 [0.706 to 0.743]
  cycle4 | 0.704 [0.681 to 0.726] | 0.700 [0.678 to 0.721]
  cycle5 | 0.679 [0.653 to 0.705] | 0.675 [0.650 to 0.700]
  cycle6 | 0.654 [0.625 to 0.684] | 0.651 [0.622 to 0.679]

5. Secondary Outcome: Health-related Quality of Life and Utility Values as Measured by EQ-5D - VAS
Description: Participants indicated on a scale of 0 (worst) to 100 (best) how good or bad their health state was on that particular day.
Time Frame: The EQ-5D VAS was administered at the beginning of the visit prior to seeing the investigator. Questionnaires were to be completed every 6 weeks (Day 1 of each cycle) for subsequent cycles and at the end of treatment visit.
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Scores on a scale
  cycle1 | 74.397 [73.219 to 75.576] | 74.656 [73.504 to 75.808]
  cycle2 | 72.649 [71.420 to 73.877] | 72.907 [71.735 to 74.080]
  cycle3 | 70.900 [69.518 to 72.281] | 71.158 [69.854 to 72.462]
  cycle4 | 69.151 [67.542 to 70.759] | 69.409 [67.891 to 70.927]
  cycle5 | 67.402 [65.520 to 69.283] | 67.660 [65.875 to 69.445]
  cycle6 | 65.653 [63.468 to 67.837] | 65.911 [63.827 to 67.996]

6. Other Pre Specified Outcome: Duration of Response
Description: Duration of response - RECIST: number of days from the date that CR or PR is first documented to date that PD is first objectively documented or to death before progression. Note: the relevant date is that of the first documentation, not the confirmation date (if participant progressed or died then censored=no) or to last observation if participant did not progress or die then censored=yes note: this last observation date should be the same as that used for time to progression.
Time Frame: From randomization of the first participant until 34 months later (cut-off date), assessed every 6 weeks
Population: The full analysis set (FAS), which was defined as all randomized participants. Duration of response was evaluated in the 14 participants in the sorafenib + placebo group and 24 participants in the sorafenib + erlotinib group who achieved their confirmed best response as CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 24 | 14
Days | 297 [100 to 427] | 168 [90 to NA] — upper bound of the confidence interval is not available due to censored data.

7. Other Pre Specified Outcome: Time to Response
Description: Time to response was the number of days from randomization to the date the CR or PR was documented (with confirmation) (Note: the relevant date is that of the first documentation, not the confirmation date).
Time Frame: From randomization of the first participant until 34 months later (cut-off date), assessed every 6 weeks
Population: The full analysis set (FAS), which was defined as all randomized participants. Time to response was evaluated in the 14 participants in the sorafenib + placebo group and 24 participants in the sorafenib + erlotinib group who achieved their confirmed best response as CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 24 | 14
Days | 84.5 [47 to 122] | 83.5 [39 to 331]

8. Other Pre Specified Outcome: Tumor Response
Description: Tumor response was the proportion of participants with the best tumor response (ie, achieving either a confirmed complete response [CR] or partial response [PR], according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria).
Time Frame: From randomization of the first participant until 34 months later (cut-off date), assessed every 6 weeks
Population: The full analysis set (FAS), which was defined as all randomized participants
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY 43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY 43-9006) + Placebo
Number analyzed (Participants) | 362 | 358
Participants | 24 | 14

ADVERSE EVENTS:
Time Frame: From start of treatment up to 30 days after the last dose of study medication
Description: ALT: alanine transaminase; AST: aspartate transaminase; CPK: creatine phosphokinase; GI: gastrointestinal; INR: international normalized ratio
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) | Sorafenib (Nexavar, BAY43-9006) + Placebo
Serious Adverse Events (participants affected / at risk) | 214/362 | 198/355
Other Adverse Events (participants affected / at risk) | 353/362 | 349/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) (N=362) | Sorafenib (Nexavar, BAY43-9006) + Placebo (N=355)
Blood - Other (Blood and lymphatic system disorders) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 1 | 4
Hemoglobin (Blood and lymphatic system disorders) | 8 | 9
INR (Blood and lymphatic system disorders) | 1 | 0
Neutrophils (Blood and lymphatic system disorders) | 0 | 1
Platelets (Blood and lymphatic system disorders) | 1 | 2
Cardiac general - Other (Cardiac disorders) | 0 | 3
Cardiac ischemia/infarction (Cardiac disorders) | 3 | 3
Conduction abnormality, asystole (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 2
Hypotension (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Pulmonary hypertension (Cardiac disorders) | 0 | 1
Supraventricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, Sinus bradycardia (Cardiac disorders) | 1 | 1
Supraventricular arrhythmia, Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia, Bigeminy (Cardiac disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Ocular - Other (Eye disorders) | 0 | 2
Uveitis (Eye disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 4 | 1
Ascites (Gastrointestinal disorders) | 15 | 13
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 12 | 5
Diarrhea (Gastrointestinal disorders) | 15 | 3
Distension (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Fistula, GI, Abdomen NOS (Gastrointestinal disorders) | 0 | 2
Fistula, GI, Anus (Gastrointestinal disorders) | 0 | 1
Fistula, GI, Stomach (Gastrointestinal disorders) | 0 | 1
GI - Other (Gastrointestinal disorders) | 1 | 4
Gastritis (Gastrointestinal disorders) | 1 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Mucositis (clinical exam), Large bowel (Gastrointestinal disorders) | 1 | 0
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Necrosis, GI, Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 | 1
Obstruction, GI, Colon (Gastrointestinal disorders) | 0 | 1
Obstruction, GI, Gallbladder (Gastrointestinal disorders) | 1 | 0
Perforation, GI, Colon (Gastrointestinal disorders) | 1 | 0
Perforation, GI, Duodenum (Gastrointestinal disorders) | 0 | 1
Perforation, GI, Stomach (Gastrointestinal disorders) | 1 | 0
Stricture, GI, Biliary tree (Gastrointestinal disorders) | 1 | 0
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1 | 1
Ulcer, GI, Esophagus (Gastrointestinal disorders) | 1 | 0
Ulcer, GI, Stomach (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Constitutional symptoms - Other (General disorders) | 13 | 20
Death not associated with CTCAE term, Death NOS (General disorders) | 6 | 1
Death not associated with CTCAE term, Disease progression NOS (General disorders) | 23 | 24
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 5 | 4
Fatigue (General disorders) | 10 | 8
Fever (General disorders) | 12 | 10
Flu-like syndrome (General disorders) | 0 | 1
No code in CTCAE (General disorders) | 3 | 10
Pain, Abdomen NOS (General disorders) | 13 | 16
Pain, Back (General disorders) | 0 | 3
Pain, Bone (General disorders) | 1 | 2
Pain, Chest wall (General disorders) | 5 | 0
Pain, Chest/Thorax NOS (General disorders) | 1 | 1
Pain, Extremity - limb (General disorders) | 1 | 0
Pain, Joint (General disorders) | 1 | 1
Pain, Muscle (General disorders) | 0 | 1
Pain, Other (General disorders) | 1 | 0
Pain, Pain NOS (General disorders) | 2 | 0
Pain, Scrotum (General disorders) | 0 | 1
Pain, Stomach (General disorders) | 4 | 0
Pain, Tumor pain (General disorders) | 1 | 1
Weight gain (General disorders) | 1 | 0
Weight loss (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary - Other (Hepatobiliary disorders) | 3 | 7
Liver dysfunction (Hepatobiliary disorders) | 35 | 32
Pancreatitis (Hepatobiliary disorders) | 1 | 2
Colitis, infectious (Infections and infestations) | 3 | 0
Infection (Documented clinically), Biliary tree (Infections and infestations) | 1 | 0
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 0 | 1
Infection (Documented clinically), Blood (Infections and infestations) | 0 | 2
Infection (Documented clinically), Lung (Pneumonia) (Infections and infestations) | 1 | 1
Infection (Documented clinically), Peritoneal cavity (Infections and infestations) | 0 | 1
Infection - Other (Infections and infestations) | 4 | 7
Infection with normal ANC, Abdomen NOS (Infections and infestations) | 1 | 1
Infection with normal ANC, Anal/perianal (Infections and infestations) | 1 | 0
Infection with normal ANC, Blood (Infections and infestations) | 3 | 3
Infection with normal ANC, Bronchus (Infections and infestations) | 1 | 0
Infection with normal ANC, Catheter-related (Infections and infestations) | 0 | 1
Infection with normal ANC, Heart (Endocarditis) (Infections and infestations) | 0 | 1
Infection with normal ANC, Kidney (Infections and infestations) | 0 | 1
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 4 | 3
Infection with normal ANC, Penis (Infections and infestations) | 0 | 1
Infection with normal ANC, Peritoneal cavity (Infections and infestations) | 1 | 1
Infection with normal ANC, Skin (cellulitis) (Infections and infestations) | 1 | 3
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 1 | 1
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC, Abdomen NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC, Anal/perianal (Infections and infestations) | 0 | 1
Infection with unknown ANC, Biliary tree (Infections and infestations) | 0 | 1
Infection with unknown ANC, Blood (Infections and infestations) | 1 | 1
Infection with unknown ANC, Cornea (Infections and infestations) | 0 | 1
Infection with unknown ANC, Duodenum (Infections and infestations) | 0 | 1
Infection with unknown ANC, Lung (Pneumonia) (Infections and infestations) | 3 | 2
Infection with unknown ANC, Peritoneal cavity (Infections and infestations) | 0 | 2
Viral hepatitis (Infections and infestations) | 1 | 0
Intraop injury, Lung (Injury, poisoning and procedural complications) | 1 | 0
ALT (Metabolism and nutrition disorders) | 3 | 0
AST (Metabolism and nutrition disorders) | 6 | 2
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 12 | 6
CPK (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 | 2
Secondary malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 1 | 6
Encephalopathy (Nervous system disorders) | 4 | 6
Mood Alteration, Agitation (Nervous system disorders) | 0 | 1
Mood alteration, Depression (Nervous system disorders) | 1 | 0
Neurology - Other (Nervous system disorders) | 0 | 1
Neuropathy: Cranial, CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 0 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 1
Neuropathy: sensory (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 2 | 3
Syncope (Fainting) (Nervous system disorders) | 2 | 3
Renal - Other (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 10 | 8
Urinary retention (Renal and urinary disorders) | 4 | 0
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 0
Bruising (Skin and subcutaneous tissue disorders) | 1 | 0
Burn (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 | 3
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
CNS hemorrhage (Vascular disorders) | 3 | 2
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage - Other (Vascular disorders) | 1 | 4
Hemorrhage pulmonary, Bronchopulmonary NOS (Vascular disorders) | 1 | 0
Hemorrhage pulmonary, Nose (Vascular disorders) | 2 | 0
Hemorrhage pulmonary, Respiratory tract NOS (Vascular disorders) | 0 | 1
Hemorrhage with surgery (Vascular disorders) | 1 | 0
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 3 | 8
Hemorrhage, GI, Anus (Vascular disorders) | 1 | 1
Hemorrhage, GI, Colon (Vascular disorders) | 2 | 0
Hemorrhage, GI, Duodenum (Vascular disorders) | 1 | 2
Hemorrhage, GI, Esophagus (Vascular disorders) | 4 | 4
Hemorrhage, GI, Liver (Vascular disorders) | 2 | 0
Hemorrhage, GI, Lower GI NOS (Vascular disorders) | 1 | 2
Hemorrhage, GI, Oral cavity (Vascular disorders) | 1 | 0
Hemorrhage, GI, Stomach (Vascular disorders) | 6 | 4
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 11 | 8
Hemorrhage, GI, Varices (Esophageal) (Vascular disorders) | 6 | 12
Hemorrhage, GI, Varices (rectal) (Vascular disorders) | 0 | 1
Hemorrhage, GU, Urinary NOS (Vascular disorders) | 1 | 0
Peripheral arterial ischemia (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 2 | 0
Thrombosis/Embolism (vascular access) (Vascular disorders) | 1 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 | 5
Vascular - Other (Vascular disorders) | 1 | 0
Visceral arterial ischemia (Vascular disorders) | 0 | 1
Blood - Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Edema: Limb (Blood and lymphatic system disorders) | 1 (1) | 4 (6)
Hemoglobin (Blood and lymphatic system disorders) | 8 (12) | 9 (15)
INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cardiac General - Other (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac ischemia/infarction (Cardiac disorders) | 3 (3) | 4 (4)
Conduction abnormality, asystole (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 3 (3) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 0 (0) | 1 (1)
SupraVentricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
SupraVentricular arrhythmia, Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
SupraVentricular arrhythmia, Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia, Bigeminy (Cardiac disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Ocular - Other (Eye disorders) | 0 (0) | 2 (3)
Uveitis (Eye disorders) | 1 (3) | 0 (0)
Anorexia (Gastrointestinal disorders) | 4 (8) | 1 (1)
Ascites (Gastrointestinal disorders) | 14 (26) | 13 (21)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 12 (14) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 15 (16) | 3 (4)
Distension (Gastrointestinal disorders) | 2 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula, GI, Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 2 (4)
Fistula, GI, Anus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fistula, GI, Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI - Other (Gastrointestinal disorders) | 1 (1) | 4 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Heartburn (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mucositis (clinical exam), Large bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrosis, GI, Colon/cecum/appendix (Gastrointestinal disorders) | 0 (0) | 1 (2)
Obstruction, GI, Colon (Gastrointestinal disorders) | 0 (0) | 1 (2)
Obstruction, GI, Gallbladder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI, Colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perforation, GI, Duodenum (Gastrointestinal disorders) | 0 (0) | 1 (2)
Perforation, GI, Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stricture, GI, Biliary tree (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1 (5) | 1 (1)
Ulcer, GI, Stomach (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constitutional Symptoms - Other (General disorders) | 11 (15) | 19 (23)
Death not associated with CTCAE term, Death NOS (General disorders) | 7 (7) | 1 (1)
Death not associated with CTCAE term, Disease Progression NOS (General disorders) | 18 (18) | 17 (17)
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 11 (14) | 8 (15)
Fever (General disorders) | 12 (15) | 11 (13)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
No Code In CTCAE (General disorders) | 3 (3) | 10 (11)
Pain, Abdomen NOS (General disorders) | 12 (19) | 15 (15)
Pain, Back (General disorders) | 0 (0) | 3 (3)
Pain, Bone (General disorders) | 1 (1) | 2 (2)
Pain, Chest wall (General disorders) | 5 (6) | 0 (0)
Pain, Chest/thorax NOS (General disorders) | 1 (1) | 1 (1)
Pain, Extremity - limb (General disorders) | 1 (1) | 0 (0)
Pain, Joint (General disorders) | 1 (1) | 1 (1)
Pain, Muscle (General disorders) | 0 (0) | 1 (1)
Pain, Other (Specify) (General disorders) | 1 (1) | 0 (0)
Pain, Pain NOS (General disorders) | 2 (2) | 0 (0)
Pain, Scrotum (General disorders) | 0 (0) | 1 (1)
Pain, Stomach (General disorders) | 4 (4) | 0 (0)
Pain, Tumor pain (General disorders) | 1 (1) | 1 (2)
Syndromes - Other (General disorders) | 0 (0) | 1 (2)
Weight gain (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary - Other (Hepatobiliary disorders) | 3 (4) | 8 (9)
Liver dysfunction (Hepatobiliary disorders) | 36 (44) | 30 (37)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Colitis, infectious (Infections and infestations) | 3 (4) | 0 (0)
Infection (Documented clinically), Biliary tree (Infections and infestations) | 1 (1) | 0 (0)
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection (Documented clinically), Blood (Infections and infestations) | 0 (0) | 2 (2)
Infection (Documented clinically), Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Infection (Documented clinically), Peritoneal Cavity (Infections and infestations) | 0 (0) | 1 (2)
Infection (Documented clinically), Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (Infections and infestations) | 5 (5) | 7 (7)
Infection with normal ANC, Abdomen NOS (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC, Anal/perianal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC, Blood (Infections and infestations) | 3 (3) | 3 (3)
Infection with normal ANC, Bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC, Catheter-related (Infections and infestations) | 0 (0) | 1 (2)
Infection with normal ANC, Heart (Endocarditis) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC, Kidney (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC, Lung (pneumonia) (Infections and infestations) | 4 (4) | 1 (1)
Infection with normal ANC, Penis (Infections and infestations) | 0 (0) | 1 (2)
Infection with normal ANC, Peritoneal cavity (Infections and infestations) | 1 (1) | 1 (2)
Infection with normal ANC, Skin (cellulitis) (Infections and infestations) | 1 (1) | 3 (6)
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC, Abdomen NOS (Infections and infestations) | 1 (2) | 0 (0)
Infection with unknown ANC, Anal/perianal (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC, Biliary tree (Infections and infestations) | 0 (0) | 1 (2)
Infection with unknown ANC, Blood (Infections and infestations) | 1 (1) | 1 (2)
Infection with unknown ANC, Cornea (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC, Duodenum (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC, Lung (pneumonia) (Infections and infestations) | 3 (3) | 2 (3)
Infection with unknown ANC, Peritoneal Cavity (Infections and infestations) | 0 (0) | 2 (2)
Viral hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Intraop injury, Lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALT (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
AST (Metabolism and nutrition disorders) | 6 (7) | 2 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 12 (20) | 5 (9)
CPK (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 2 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 6 (9) | 0 (0)
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Secondary Malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 2 (5)
CNS ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 6 (9)
Encephalopathy (Nervous system disorders) | 4 (16) | 6 (8)
Mood Alteration, Agitation (Nervous system disorders) | 0 (0) | 1 (1)
Mood Alteration, Depression (Nervous system disorders) | 1 (3) | 0 (0)
Neurology - Other (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: Cranial, CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 0 (0) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 1 (14) | 1 (3)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 2 (6)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 3 (4)
Renal - Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 10 (12) | 8 (13)
Urinary retention (Renal and urinary disorders) | 4 (5) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 7 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (4)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
CNS hemorrhage (Vascular disorders) | 3 (4) | 2 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (2)
Hemorrhage - Other (Vascular disorders) | 1 (1) | 4 (5)
Hemorrhage pulmonary, Bronchopulmonary NOS (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage pulmonary, Nose (Vascular disorders) | 2 (2) | 0 (0)
Hemorrhage pulmonary, Respiratory tract NOS (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage with surgery (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 3 (3) | 8 (10)
Hemorrhage, GI, Anus (Vascular disorders) | 1 (1) | 1 (1)
Hemorrhage, GI, Colon (Vascular disorders) | 2 (2) | 0 (0)
Hemorrhage, GI, Duodenum (Vascular disorders) | 1 (1) | 2 (2)
Hemorrhage, GI, Esophagus (Vascular disorders) | 4 (7) | 4 (4)
Hemorrhage, GI, Liver (Vascular disorders) | 2 (2) | 1 (1)
Hemorrhage, GI, Lower GI NOS (Vascular disorders) | 1 (1) | 1 (3)
Hemorrhage, GI, Oral cavity (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage, GI, Stomach (Vascular disorders) | 6 (7) | 4 (4)
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 11 (13) | 7 (9)
Hemorrhage, GI, Varices (esophageal) (Vascular disorders) | 6 (7) | 11 (18)
Hemorrhage, GI, Varices (rectal) (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage, GU, Urinary NOS (Vascular disorders) | 1 (2) | 0 (0)
Peripheral arterial ischemia (Vascular disorders) | 0 (0) | 2 (3)
Phlebitis (Vascular disorders) | 2 (3) | 0 (0)
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (7) | 5 (11)
Vascular - Other (Vascular disorders) | 1 (2) | 0 (0)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Erlotinib (Tarceva) (N=362) | Sorafenib (Nexavar, BAY43-9006) + Placebo (N=355)
Edema: Limb (Blood and lymphatic system disorders) | 83 | 76
Hemoglobin (Blood and lymphatic system disorders) | 67 | 53
INR (Blood and lymphatic system disorders) | 19 | 19
Leukocytes (Blood and lymphatic system disorders) | 16 | 21
Platelets (Blood and lymphatic system disorders) | 44 | 51
Hypertension (Cardiac disorders) | 71 | 86
Anorexia (Gastrointestinal disorders) | 156 | 135
Ascites (Gastrointestinal disorders) | 77 | 91
Constipation (Gastrointestinal disorders) | 51 | 76
Dehydration (Gastrointestinal disorders) | 21 | 8
Diarrhea (Gastrointestinal disorders) | 272 | 211
Distension (Gastrointestinal disorders) | 26 | 24
Dry mouth (Gastrointestinal disorders) | 14 | 24
Flatulence (Gastrointestinal disorders) | 24 | 19
GI - Other (Gastrointestinal disorders) | 31 | 30
Gastritis (Gastrointestinal disorders) | 26 | 12
Heartburn (Gastrointestinal disorders) | 30 | 22
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 72 | 53
Nausea (Gastrointestinal disorders) | 91 | 113
Taste Alteration (Gastrointestinal disorders) | 20 | 10
Vomiting (Gastrointestinal disorders) | 81 | 80
Constitutional symptoms - Other (General disorders) | 20 | 25
Fatigue (General disorders) | 183 | 191
Fever (General disorders) | 71 | 64
Insomnia (General disorders) | 38 | 44
Pain, Abdomen NOS (General disorders) | 115 | 120
Pain, Back (General disorders) | 41 | 48
Pain, Chest/Thorax NOS (General disorders) | 10 | 24
Pain, Extremity - limb (General disorders) | 14 | 23
Pain, Head/Headache (General disorders) | 32 | 51
Pain, Joint (General disorders) | 24 | 18
Pain, Muscle (General disorders) | 21 | 20
Pain, Other (General disorders) | 19 | 22
Weight loss (General disorders) | 127 | 109
Liver dysfunction (Hepatobiliary disorders) | 23 | 21
Infection - Other (Infections and infestations) | 14 | 25
ALT (Metabolism and nutrition disorders) | 44 | 43
AST (Metabolism and nutrition disorders) | 78 | 75
Alkaline phosphatase (Metabolism and nutrition disorders) | 23 | 26
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 62 | 74
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 24
Hypokalemia (Metabolism and nutrition disorders) | 32 | 21
Hyponatremia (Metabolism and nutrition disorders) | 17 | 21
Hypophosphatemia (Metabolism and nutrition disorders) | 40 | 39
Lipase (Metabolism and nutrition disorders) | 20 | 13
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 27 | 21
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 26 | 28
Dizziness (Nervous system disorders) | 18 | 25
Mood alteration, Depression (Nervous system disorders) | 15 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 60
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 34 | 38
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Voice changes (Respiratory, thoracic and mediastinal disorders) | 31 | 30
Acne (Skin and subcutaneous tissue disorders) | 53 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 46 | 84
Dermatology - Other (Skin and subcutaneous tissue disorders) | 54 | 39
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 34
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 136 | 169
Pruritus (Skin and subcutaneous tissue disorders) | 43 | 46
Rash/desquamation (Skin and subcutaneous tissue disorders) | 187 | 143
Hemorrhage pulmonary, Nose (Vascular disorders) | 65 | 25
Edema: Limb (Blood and lymphatic system disorders) | 82 (176) | 74 (150)
Hemoglobin (Blood and lymphatic system disorders) | 65 (200) | 49 (129)
INR (Blood and lymphatic system disorders) | 19 (36) | 18 (56)
Leukocytes (Blood and lymphatic system disorders) | 17 (48) | 20 (41)
Platelets (Blood and lymphatic system disorders) | 45 (156) | 50 (186)
Hypertension (Cardiac disorders) | 72 (339) | 86 (336)
Anorexia (Gastrointestinal disorders) | 153 (479) | 135 (383)
Ascites (Gastrointestinal disorders) | 76 (192) | 86 (205)
Constipation (Gastrointestinal disorders) | 46 (77) | 72 (145)
Dehydration (Gastrointestinal disorders) | 21 (30) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 273 (1079) | 211 (784)
Distension (Gastrointestinal disorders) | 26 (98) | 22 (61)
Dry mouth (Gastrointestinal disorders) | 13 (33) | 24 (105)
Flatulence (Gastrointestinal disorders) | 24 (63) | 19 (51)
GI - Other (Gastrointestinal disorders) | 31 (120) | 29 (81)
Gastritis (Gastrointestinal disorders) | 24 (53) | 13 (32)
Heartburn (Gastrointestinal disorders) | 28 (111) | 21 (47)
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 72 (176) | 53 (134)
Nausea (Gastrointestinal disorders) | 90 (212) | 109 (259)
Taste Alteration (Gastrointestinal disorders) | 20 (82) | 10 (33)
Vomiting (Gastrointestinal disorders) | 82 (140) | 78 (150)
Constitutional Symptoms - Other (General disorders) | 21 (33) | 25 (53)
Fatigue (General disorders) | 184 (676) | 192 (779)
Fever (General disorders) | 71 (112) | 64 (107)
Insomnia (General disorders) | 36 (151) | 43 (105)
Pain, Abdomen NOS (General disorders) | 112 (339) | 112 (312)
Pain, Back (General disorders) | 40 (132) | 48 (110)
Pain, Chest/thorax NOS (General disorders) | 10 (15) | 25 (47)
Pain, Extremity - limb (General disorders) | 15 (46) | 23 (74)
Pain, Head/headache (General disorders) | 31 (60) | 51 (117)
Pain, Joint (General disorders) | 24 (56) | 19 (48)
Pain, Muscle (General disorders) | 21 (78) | 19 (54)
Pain, Other (Specify) (General disorders) | 20 (28) | 25 (51)
Weight loss (General disorders) | 127 (552) | 111 (465)
Liver dysfunction (Hepatobiliary disorders) | 21 (35) | 21 (39)
Infection - Other (Infections and infestations) | 12 (19) | 25 (43)
ALT (Metabolism and nutrition disorders) | 43 (159) | 39 (92)
AST (Metabolism and nutrition disorders) | 76 (259) | 74 (217)
Alkaline phosphatase (Metabolism and nutrition disorders) | 19 (67) | 24 (66)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 59 (131) | 74 (166)
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 (50) | 27 (50)
Hypocalcemia (Metabolism and nutrition disorders) | 21 (66) | 24 (67)
Hypokalemia (Metabolism and nutrition disorders) | 31 (64) | 21 (41)
Hyponatremia (Metabolism and nutrition disorders) | 18 (22) | 21 (35)
Hypophosphatemia (Metabolism and nutrition disorders) | 39 (135) | 38 (89)
Lipase (Metabolism and nutrition disorders) | 20 (57) | 13 (24)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 26 (52) | 20 (53)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 25 (92) | 28 (139)
Dizziness (Nervous system disorders) | 18 (52) | 25 (45)
Mood Alteration, Depression (Nervous system disorders) | 15 (35) | 23 (119)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (138) | 60 (111)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 35 (79) | 40 (74)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 13 (32) | 20 (41)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 31 (120) | 31 (116)
Acne (Skin and subcutaneous tissue disorders) | 53 (210) | 13 (46)
Alopecia (Skin and subcutaneous tissue disorders) | 46 (222) | 84 (352)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 55 (184) | 39 (142)
Dry skin (Skin and subcutaneous tissue disorders) | 36 (122) | 33 (114)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 136 (723) | 169 (805)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (83) | 44 (101)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 186 (785) | 141 (536)
Hemorrhage pulmonary, Nose (Vascular disorders) | 63 (123) | 25 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must send a draft manuscript of the publication or abstract to the sponsor 30 days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.